CLINICAL TRIAL: NCT02850939
Title: Improving Adherence to Endocrine Hormonal Therapy Among Breast Cancer Patients
Brief Title: Improving Adherence to EHT Among Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HSC20160245H
Record Dates: First submitted 2016-07-20; First posted 2016-08-01 (Estimated); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Endocrine hormonal therapy; mHealth
MeSH Terms: conditions — Breast Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile phone app + patient navigation (Experimental): Patients assigned to the intervention group (60) will: 1) use the personalized mobile phone app in their preferred language for a duration of 6 months; and 2) receive assistance from a patient navigator. They will also continue to receive the usual EHT care provided at the MCC's breast clinic.
  Interventions: Behavioral: Mobile phone app + patient navigation
- Usual care (No Intervention): Patients assigned to the control (usual care) group (60) will receive the usual EHT care and materials offered at the MCC's breast clinic.

INTERVENTIONS:
Behavioral: Mobile phone app + patient navigation — The intervention group will receive two components: 1) a culturally sensitive, personalized and easy to use smartphone app; and 2) support from a patient navigator. The intervention is based in Social Cognitive Theory and principles of motivational interviewing - and will feature basic components of individual empowerment, motivation and engagement, including knowledge, attitudes, skills, peer modeling, social support/reinforcement and self-efficacy beliefs and expectations
  Arms: Mobile phone app + patient navigation

SUMMARY:
Adjuvant endocrine hormonal therapy (EHT) is highly effective and appropriate for nearly all breast cancer patients with hormone receptor-positive tumors, which represent 75% of all breast cancer diagnoses. Long-term use of EHT reduces cancer recurrence rates and cuts the risk of death nearly in half during the second decade after diagnosis, research shows. Despite the proven benefits, about 33% of women who are prescribed EHT do not take their medication as prescribed (less than 80% take their daily dosage) and are thus at higher risk of recurrence and death.

This educational randomized controlled study will develop and pilot-test a bilingual, culturally tailored, personalized, interactive mobile application (app) in combination with patient navigation to promote and improve adherence to endocrine hormonal therapy (EHT) among breast cancer patients.

DETAILED DESCRIPTION:
The proposed two-year study involves a 2-group randomized control trial with 3-time assessments (baseline, 3 and 6 months) and will enroll 120 breast cancer patients who are prescribed EHT and are attending the breast clinic at the Mays Cancer Center (MCC), a National Cancer Institute-designated cancer center at the University of Texas Health Science Center at San Antonio. The intervention group will receive two components: 1) a bilingual, culturally tailored, personalized, interactive mobile app; and 2) support from a patient navigator. The control group will receive the usual care and information provided by the MCC's breast clinic and pharmacy to patients undergoing oral EHT. The intervention components are based in Social Cognitive Theory and elements of Motivational Interviewing.

The proposed study aims to:

1. Develop a bilingual, culturally tailored, personalized, interactive mobile application (app) to promote and improve EHT adherence among breast cancer patients diagnosed with hormone receptor-positive breast cancer. The app will empower patients' self-monitoring and management, as well as facilitate patient education, early identification and reporting of side effects, delivery of self-care advice, and timely feedback through direct interaction between the patient and the oncology team when necessary.
2. Conduct a 2-group randomized controlled study to assess the feasibility and effectiveness of a bilingual, culturally tailored, personalized, interactive app + patient navigation (PN) to promote EHT adherence compared to usual care among patients diagnosed with hormone receptor-positive breast cancer and who are prescribed EHT.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking adult patients, 18 years of age and older who: a) are diagnosed with hormone receptor-positive breast cancer and prescribed endocrine hormonal treatment (EHT); b) own a cell phone, are able to send and receive text message and access the internet; and c) are able to provide informed consent to participate in the study.

Exclusion Criteria:

* Patients who: (a) are unable to provide consent due to a mental, emotional, or physical handicap, that keep them from understanding the consent information; (b) do not own a smart phone; (c) are unable to respond to text messages and questions or unable download the study app; d) are unable to see the app and study materials and videos (i.e., are blind, deaf)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in Adherence to EHT | Outcome will be assessed at 3 points: baseline, 3 and 6 months
  We will review prescribing and refill records for EHT (tamoxifen or aromatase inhibitors -AIs) and the number of days cover by each prescription, the number of dispensed tablets and the daily dose, to calculate an adherence index across the 6-month intervention.18 In addition we will use monthly self-reporting data via the mobile app using 3 questions developed by the research team.

SECONDARY OUTCOMES:
Change in Quality of Life | Outcome will be assessed at 3 points: baseline, 3 and 6 months
  Quality of life will be measured by the Functional Assessment of Cancer Therapy-General (FACT-G) questionnaire. This questionnaire is well validated and has been used in multiple studies around the world.
Change in Anxiety | Outcome will be assessed at 3 points: baseline, 3 and 6 months
  To assess anxiety we will use the Generalized Anxiety Disorder 7-item scale (GAD-7), a validated tool used in clinical practice and research studies to assess the severity of anxiety.
Usability and satisfaction with the mobile app | Outcome will be measured at 6 months
  we will assess usability and satisfaction of the mobile app by including a small set of questions developed by the research team with response options ranging from completely agree to completely disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Amelie G. Ramirez, DrPH, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Mays Cancer Center - MCC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data won't be shared as per protocol. Results will be presented in aggregated form without any identifiers.

REFERENCES:
- [Background] Chalela P, Munoz E, Inupakutika D, Kaghyan S, Akopian D, Kaklamani V, Lathrop K, Ramirez A. Improving adherence to endocrine hormonal therapy among breast cancer patients: Study protocol for a randomized controlled trial. Contemp Clin Trials Commun. 2018 Oct 17;12:109-115. doi: 10.1016/j.conctc.2018.10.001. eCollection 2018 Dec. PMID 30377674